CLINICAL TRIAL: NCT01803113
Title: Sofia hCG FIA Field Study
Status: Completed | Type: Observational
Sponsor: Quidel Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-0144-01
Record Dates: First submitted 2013-02-21; First posted 2013-03-04 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Pregnancy, Early Detection
Keywords: Pregnancy; hCG

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Leftover urine specimens may be retained to be used for further product testing.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Sofia hCG FIA — Qualitative detection via immunofluorescence technology of increased level of hCG present in urine.

SUMMARY:
The objective of this field study is to demonstrate the clinical performance of the Sofia hCG FIA Test, using urine specimens from females of childbearing age.

DETAILED DESCRIPTION:
Subjects presenting for pregnancy testing will provide urine specimens that will be tested with the Sofia hCG FIA test and the comparator pregnancy test that will detect levels of hCG of 20mIU as positive for pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects of childbearing age, who are being screened for pregnancy and who have signed the informed consent

Exclusion Criteria:

* Subject is post-menopausal.
* Subject within the past six weeks has experienced any of the following: delivered a newborn; had an abortion or a natural termination (miscarriage); or, received hCG supplements.
* Subject has had a hysterectomy.
* Unable to understand and consent to participation.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any female of childbearing potential being screened for pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 975 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Determination of presence of hCG in urine | 1 day
  Clinical performance will be based on comparison of Sofia hCG FIA test results to those obtained from an FDA-cleared hCG test.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Jose Castaneda, MD, Boynton Beach, Florida
  - NECCR of Massachusetts, LLC, Fall River, Massachusetts
  - New England Center for Clinical Research Fall River,LLC (NECCR), Fall River, Massachusetts
  - Partners In Obstetrics and Gynecology, Inc., Pawtucket, Rhode Island
  - Planned Parenthood Gulf Coast, Houston, Texas